CLINICAL TRIAL: NCT03480646
Title: A Phase 1b/2 Study of CPI-1205, a Small Molecule Inhibitor of EZH2, Combined With Enzalutamide or Abiraterone/Prednisone in Patients With Metastatic Castration Resistant Prostate Cancer
Brief Title: ProSTAR: A Study Evaluating CPI-1205 in Patients With Metastatic Castration Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Constellation Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1205-201
Record Dates: First submitted 2018-03-07; First posted 2018-03-29 (Actual); Results first posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Castration Resistant Prostate Cancer (mCRPC)
Keywords: Phase 1/2; Oncology; EZH2 Inhibitor
MeSH Terms: conditions — Neoplasms | interventions — (R)-N-((4-methoxy-6-methyl-2-oxo-1,2-dihydropyridin-3-yl)methyl)-2-methyl-1-(1-(1-(2,2,2-trifluoroethyl)piperidin-4-yl)ethyl)-1H-indole-3-carboxamide; Cobicistat; enzalutamide; abiraterone; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Phase 1b Dose Escalation: CPI-1205 400 mg BID + Cobi + Enza (Experimental): CPI-1205 400 mg BID in combination with Cobicistat 150 mg PO BID and Enzalutamide 160 mg PO QD (28-day cycles)
  Interventions: Drug: CPI-1205; Drug: Cobicistat; Drug: Enzalutamide
- Phase 1b Dose Escalation: CPI-1205 400 mg BID + Cobi+ Abi/Pred (Experimental): CPI-1205 400 mg BID in combination with Cobicistat 150 mg PO BID and Abiraterone 100 mg PO QD and Prednisone 5 mg PO BID (28-day cycle)
  Interventions: Drug: CPI-1205; Drug: Cobicistat; Drug: Abiraterone; Drug: Prednisone
- Phase 1b Dose Escalation: CPI-1205 800 mg TID + Enza (Experimental): CPI-1205 800 mg TID in combination with Enzalutamide 160 mg PO QD (28-day cycle)
  Interventions: Drug: CPI-1205; Drug: Enzalutamide
- Phase 1b Dose Escalation: CPI-1205 800 mg TID + Abi/Pred (Experimental): CPI-1205 800 mg TID in combination with Abiraterone 100 mg PO QD and Prednisone 5 mg PO BID (28-day cycle)
  Interventions: Drug: CPI-1205; Drug: Abiraterone; Drug: Prednisone
- Phase 1b HPEC: CPI-1205 800 mg TID + Enza (Experimental): CPI-1205 800 mg TID highly pretreated expansion cohort (HEPC) in combination with Enzalutamide 160 mg PO QD (28-day cycles)
  Interventions: Drug: CPI-1205; Drug: Enzalutamide
- Phase 2 Randomized Controlled Group: Enza (Active Comparator): Drug: Enzalutamide 160mg PO QD (28-day cycles)
  Interventions: Drug: Enzalutamide
- Phase 2 Randomized at RP2D: CPI-1205 800 mg TID + Enza (Experimental): CPI-1205 (at Recommended Phase 2 Dose [RP2D]) in combination with Drug: Enzalutamide 160 mg PO QD
  Interventions: Drug: CPI-1205; Drug: Enzalutamide
- Phase 2 Single Arm at RP2D: CPI-1205 800 mg TID + Abi/Pred (Experimental): CPI-1205 at 800 mg TID (Recommended Phase 2 Dose [RP2D]) 800 mg TID in combination with Abiraterone 1000 mg PO QD and Prednisone 5 mg PO BID (28-day cycles)
  Interventions: Drug: CPI-1205; Drug: Abiraterone; Drug: Prednisone

INTERVENTIONS:
Drug: CPI-1205 — CPI-1205: Either 400 mg BID or 800 mg TID during Phase 1 dose-escalation and RP2D, 800 mg TID, for Phase 2
  Arms: Phase 1b Dose Escalation: CPI-1205 400 mg BID + Cobi + Enza; Phase 1b Dose Escalation: CPI-1205 400 mg BID + Cobi+ Abi/Pred; Phase 1b Dose Escalation: CPI-1205 800 mg TID + Abi/Pred; Phase 1b Dose Escalation: CPI-1205 800 mg TID + Enza; Phase 1b HPEC: CPI-1205 800 mg TID + Enza; Phase 2 Randomized at RP2D: CPI-1205 800 mg TID + Enza; Phase 2 Single Arm at RP2D: CPI-1205 800 mg TID + Abi/Pred
Drug: Cobicistat — Cobicistat 150 mg PO BID
  Arms: Phase 1b Dose Escalation: CPI-1205 400 mg BID + Cobi + Enza; Phase 1b Dose Escalation: CPI-1205 400 mg BID + Cobi+ Abi/Pred
Drug: Enzalutamide — Enzalutamide 160mg PO QD
  Arms: Phase 1b Dose Escalation: CPI-1205 400 mg BID + Cobi + Enza; Phase 1b Dose Escalation: CPI-1205 800 mg TID + Enza; Phase 1b HPEC: CPI-1205 800 mg TID + Enza; Phase 2 Randomized Controlled Group: Enza; Phase 2 Randomized at RP2D: CPI-1205 800 mg TID + Enza
Drug: Abiraterone — Abiraterone 1000mg PO QD
  Arms: Phase 1b Dose Escalation: CPI-1205 400 mg BID + Cobi+ Abi/Pred; Phase 1b Dose Escalation: CPI-1205 800 mg TID + Abi/Pred; Phase 2 Single Arm at RP2D: CPI-1205 800 mg TID + Abi/Pred
Drug: Prednisone — Prednisone 5mg PO BID
  Arms: Phase 1b Dose Escalation: CPI-1205 400 mg BID + Cobi+ Abi/Pred; Phase 1b Dose Escalation: CPI-1205 800 mg TID + Abi/Pred; Phase 2 Single Arm at RP2D: CPI-1205 800 mg TID + Abi/Pred

SUMMARY:
This was an open-label Phase 1b/2 study involving oral administration of CPI-1205 in combination with either enzalutamide or abiraterone/prednisone in male patients with metastatic Castration-Resistant Prostate Cancer. The study was designed to determine the maximum tolerated dose (MTD) and the recommended Phase II dose (RP2D) based on the safety, tolerability, pharmacokinetic, and efficacy profiles of CPI-1205 in combination with either enzalutamide or abiraterone/prednisone.

Following the determination of the MTD and RP2D, the study proceeded to Phase 2. Patients in Phase 2 received CPI-1205 at the RP2D in combination with either enzalutamide or abiraterone/prednisone versus either enzalutamide or abiraterone/prednisone as a control arm.

DETAILED DESCRIPTION:
Study CPI-1205-201 was a Phase 1b/2, multi-center, open-label study of CPI-1205 alone and with cobicistat in subjects with mCRPC in combination with either enzalutamide or abiraterone/prednisone. The study initially had two phases: a Phase 1 dose-finding, dose-escalation study intended to establish the Recommended Phase 2 Dose (RP2D) of CPI-1205 for the Phase 2 portion.

The study underwent three amendments.

PHASE 1b In the Phase 1b dose-escalation phase and prior to Amendment 2, subjects were enrolled into Phase 1b dose level CPI-1205 PO three times daily (TID) + enzalutamide or abiraterone/prednisone.

In Amendment 2, new subjects were enrolled into cohorts including:

Dose-escalating CPI-1205 PO twice daily (BID) + fixed-dose cobicistat PO BID + enzalutamide Dose-escalating CPI-1205 PO BID + fixed-dose cobicistat PO BID + abiraterone/prednisone In Amendment 3, Phase 1b expansion cohort(s) were added in the heavily pretreated population (HPEC). An HPEC began enrollment if 0 out of 3 or 1 out of 6 subjects treated with a specific regimen (i.e., CPI-1205 with or without cobicistat, in combination with enzalutamide or abiraterone) at a given dose level during Phase 1b dose escalation experienced a dose-limiting toxicity (DLT).

Following determination of the maximum tolerated dose (MTD) in each of the CPI-1205 BID + cobicistat combinations (and possibly in the CPI-1205 TID combination) and after evaluation of the BID cohorts without cobicistat (if applicable), only one of the CPI-1205 dosing schedules was selected as the RP2D for each combination. One or both combinations proceeded to Phase 2 after consideration of pharmacokinetic (PK) and pharmacodynamic (PD) results, data from the HPEC(s), and safety data.

PHASE 2 If only one partner product was chosen for Phase 2, the study proceeded as an open-label randomized Phase 2 trial, with subjects randomized to either the combination arm (CPI-1205 at the RP2D [with or without cobicistat] in combination with enzalutamide or abiraterone/prednisone) or the control arm (enzalutamide or abiraterone/prednisone as monotherapy). If both partner products were chosen, the second Phase 2 was either a second open-label randomized trial or a single-arm Phase 2 trial (following a Simon's 2-stage design). The design of the second trial was determined by the Sponsor based on preliminary efficacy and PK.

CPI-1205 was administered orally TID or BID (as of Amendment 2). Cobicistat dosing began with one dose the evening prior to Day 1 of CPI-1205 and continued PO BID starting on Day 1. Enzalutamide and abiraterone were given PO once daily, and prednisone was given PO BID (or at the investigator's discretion).

Successive 28-day treatment cycles were repeated without planned breaks, as long as the combination was well tolerated, until radiographic disease progression, unequivocal clinical progression, or planned initiation of another systemic treatment. Investigators could continue treatment in subjects with progression in one site if other lesions might benefit. Subjects in the control arm who progressed had the option to cross over to the combination arm, provided they met eligibility criteria.

ELIGIBILITY:
PHASE 1b DOSE ESCALATION

Inclusion Criteria for Phase 1b Dose Escalation

Patients must meet all the following criteria to be enrolled in this study:

1. Age ≥ 18 years
2. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
3. Life expectancy of at least 12 weeks
4. Histologically or cytologically confirmed adenocarcinoma of the prostate (pure small cell carcinoma excluded)
5. Documented metastatic disease
6. Must have undergone bilateral orchiectomy (surgical castration) or willing to continue gonadotropin-releasing hormone (GnRH) analog or antagonist (medical castration)
7. Serum testosterone < 50 ng/dL
8. Progressive disease in the setting of medical or surgical castration (i.e., Castration-resistant Prostate Cancer [CRPC]) as assessed by the investigator and includes at least one of the following:

   1. Evidence of progression as measured by PSA increase of ≥ 25% and an absolute increase of ≥ 2 ng/mL in < 6 months from end of last therapy prior to enrollment and/or
   2. Soft tissue disease progression as per Response Evaluation Criteria in Solid Tumors (RECIST) and/or
   3. Bone disease progression defined by two or more new lesions on bone scan
9. Bisphosphonate or denosumab therapy allowed provided dose has been stable for at least 4 weeks prior to Day 1 of treatment
10. Prior treatment:

    1. Prior treatment for metastatic CRPC (mCRPC) must have included at least one line with a second-generation androgen inhibitor (e.g., abiraterone, enzalutamide, apalutamide, daralutamide)
    2. Prior chemotherapy permitted when administered in the metastatic hormone-sensitive prostate cancer setting. In addition, up to one line of chemotherapy is allowed in the mCRPC setting.
    3. Prior treatment with sipuleucel-T, radium-223, or other non-chemotherapy based treatments for mCRPC (e.g., olaparib, pembrolizumab) is allowed.
11. Recovery from recent surgery, radiotherapy, chemotherapy or other anti-cancer treatment to baseline or ≤ Grade 1 (other than alopecia)
12. Demonstrate adequate organ function as defined in the table below; all Screening labs obtained within 28 days prior to Day 1 of treatment.
13. Patients who have not undergone a bilateral orchiectomy and have a female partner of childbearing potential must use an adequate barrier method of contraception during study treatment and for 90 days after receiving the last dose of CPI-1205
14. Willing to provide access to archival tumor tissue for research purposes
15. Ability to swallow and retain oral medications
16. Ability to understand and willingness to sign an IRB approved written informed consent form (ICF) and authorization permitting release of personal health information including genetic testing relevant to cancer.
17. Able to comply with study visit schedule and assessments

Exclusion Criteria for Phase 1b Dose Escalation

Patients who meet any of the following criteria will not be enrolled in the study:

1. Known symptomatic brain metastases
2. Treatment with any of the following for prostate cancer within the indicated timeframe prior to Day 1 of treatment

   1. First generation: AR antagonists (e.g., bicalutamide, nilutamide, flutamide) within 4 weeks
   2. 5 alpha reductase inhibitors, ketoconazole, estrogens (including diethylstilbesterol [DES]), or progesterones within 2 weeks
   3. Chemotherapy within 3 weeks
   4. Biologic therapy within 4 weeks
   5. Investigational therapy within 3 weeks (or within a time interval less than at least 5 half-lives of the investigational agent [if known], whichever is longer).
   6. Immunotherapy within 4 weeks
   7. Radionuclide therapy within 4 weeks
3. Radiation therapy for the treatment of metastasis within 1 week prior to Day 1 of treatment
4. Herbal products that may decrease PSA levels within 4 weeks prior to day 1 of treatment
5. Systemic steroids greater than 10 mg of prednisone/prednisolone per day within 4 weeks prior to day 1 of treatment
6. Major surgery within 4 weeks prior to Day 1 of treatment
7. Planned palliative procedures for alleviation of bone pain such as radiation therapy or surgery
8. Structurally unstable bone lesions concerning for impending fracture
9. Clinically significant cardiovascular disease including:

   1. Myocardial infarction (MI)/Stroke within 6 months prior to Day 1 of treatment
   2. Uncontrolled angina within 3 months
   3. Congestive heart failure (CHF) with New York Heart Association (NYHA) Class 3 or 4
   4. History of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsades de pointes)
   5. Uncontrolled hypertension (systolic blood pressure (BP) > 170 mmHg or diastolic BP > 105 mmHg at screening) despite 2 concomitant antihypertensive therapies
   6. QT interval corrected by the Fridericia correction formula (QTcF) > 500 msec on the screening ECG
10. Active or symptomatic viral hepatitis or chronic liver disease
11. History of unresolved adrenal dysfunction
12. GI disorder that negatively affects absorption
13. Required treatment with one of the prohibited concomitant medications;
14. Achlorhydria, either documented or suspected on the basis of an associated disease (e.g., pernicious anemia, atrophic gastritis, or certain gastric surgical procedures)
15. History of seizure, underlying brain injury with loss of consciousness, transient ischemic attack within 12 months prior to Day 1 of treatment, cerebral vascular accident or brain arteriovenous malformation
16. Known additional malignancy that is active and/or progressive requiring treatment; exceptions include basal cell or squamous cell skin cancer, in situ bladder cancer, or other cancer for which the patient has been disease-free for at least two years
17. Any other concurrent severe and/or uncontrolled concomitant medical condition that could compromise participation in the study (e.g., clinically significant pulmonary disease, clinically significant psychiatric or neurological disorder, active or uncontrolled infection)
18. Patient unwilling or unable to comply with this study protocol

PHASE 1b: HEAVILY PRETREATED EXPANSION COHORT (HPEC)

Inclusion Criteria for Phase 1b HPEC

Patients must meet all the following criteria to be enrolled in this study:

1. Age ≥ 18 years
2. ECOG Performance Status 0-1
3. Life expectancy of at least 12 weeks
4. Histologically or cytologically confirmed adenocarcinoma of the prostate (pure small cell carcinoma excluded)
5. Documented metastatic disease
6. At least 1 measurable lymph node per Prostate Cancer Clinical Trials Working Group 3 (PCWG3)
7. Must have undergone bilateral orchiectomy (surgical castration) or willing to continue GnRH analog or antagonist (medical castration)
8. Serum testosterone < 50 ng/dL
9. Progressive disease in the setting of medical or surgical castration (i.e., CRPC) as assessed by the investigator and that includes at least 1 of the following:

   1. Evidence of progression as measured by PSA defined as: PSA at least 2 ng/mL (or PSA at least 1 ng/mL if PSA progression is the only manifestation of progressive disease) and rising PSA by at least 2 consecutive measurements a minimum of 1-week apart and/or
   2. Soft tissue disease progression as per RECIST 1.1 and/or
   3. Bone disease progression defined by two or more new lesions on bone scan
10. Prior treatment:

    1. Only 1 prior line of a second-generation androgen inhibitor from a different class than the one chosen for the applicable phase 2 study (the 2 classes are CYP17 inhibitors [e.g., abiraterone, orteronel] and AR inhibitors [e.g., enzalutamide, apalutamide]). Patient must have progressed after ≥ 24 weeks of treatment with this second generation angrogen inhibitor.
    2. The last second-generation androgen inhibitor treatment received must not be from the same class as that incorporated in the applicable HPEC; i.e., if the HPEC incorporates enzalutamide, the last second generation androgen inhibitor therapy cannot be enzalutamide, apalutamide, etc.
    3. Prior chemotherapy for mCRPC must have included at least 1 and no more than 2 prior lines of taxane-based chemotherapy administered in the metastatic hormone-sensitive prostate cancer setting is allowed
    4. Prior treatment with sipuleucel-T, radium-223, or other non-chemotherapy-based treatments for mCRPC (e.g., olaparib, pembrolizumab, nivolumab) is allowed.
11. Recovery from recent surgery, radiotherapy, chemotherapy or other anti-cancer treatment to baseline or ≤ Grade 1 (other than alopecia)
12. Demonstrate adequate organ function as defined in the table below; all Screening labs to be obtained within 28 days prior to Day 1 of treatment
13. Patients who had not undergone a bilateral orchiectomy and have a female partner of childbearing potential must use an adequate barrier method of contraception during study treatment and for 90 days after receiving the last dose of CPI-1205
14. Willing to provide access to archival tumor tissue for research purposes
15. Ability to swallow and retain oral medications
16. Ability to understand and willingness to sign an IRB approved written ICF and authorization permitting release of personal health information including genetic testing relevant to cancer.
17. Able to comply with study visit schedule and assessments

Exclusion Criteria for Phase 1b HPEC

Patients meeting any of the following criteria will not be enrolled in the study:

1. Known symptomatic brain metastases
2. Treatment with any of the following for prostate cancer within the indicated timeframe prior to Day 1 of treatment

   1. First-generation: AR antagonists (e.g., bicalutamide, nilutamide, flutamide) within 4 weeks
   2. 5-alpha reductase inhibitors, ketoconazole, estrogens (including DES), or progesterones within 2 weeks
   3. Chemotherapy within 3 weeks
   4. Biologic therapy within 4 weeks
   5. Investigational therapy within 3 weeks (or within a time interval less than at least 5 half-lives of the investigational agent [if known], whichever is longer).
   6. Immunotherapy within 4 weeks
   7. Radionuclide therapy within 4 weeks
3. Radiation therapy for the treatment of metastasis within 1 week prior to Day 1 of treatment
4. Herbal products that may decrease PSA levels within 4 weeks prior to Day 1 of treatment
5. Systemic steroids greater than 10 mg of prednisone/prednisolone per day within 4 weeks prior to Day 1 of treatment
6. Major surgery within 4 weeks prior to Day 1 of treatment
7. Structurally unstable bone lesions concerning for impending fracture
8. Clinically significant cardiovascular disease including:

   1. MI/Stroke within 6 months prior to Day 1 of treatment
   2. Uncontrolled angina within 3 months
   3. CHF with NYHA Class 3 or 4
   4. History of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsades de pointes)
   5. Uncontrolled hypertension (systolic BP > 170 mmHg or diastolic BP > 105 mmHg at screening) despite two concomitant antihypertensive therapies
   6. QTcF >500 msec on the screening ECG
9. Active or symptomatic viral hepatitis or chronic liver disease
10. History of unresolved adrenal dysfunction
11. GI disorder that negatively affects absorption
12. Required treatment with one of the prohibited concomitant medications
13. Achlorhydria, either documented or suspected on the basis of an associated disease (e.g., pernicious anemia, atrophic gastritis, or certain gastric surgical procedures)
14. History of seizure, underlying brain injury with loss of consciousness, transient ischemic attack within 12 months prior to day 1 of treatment, cerebral vascular accident or brain arteriovenous malformation
15. Known additional malignancy that is active and/or progressive requiring treatment; exceptions include basal cell or squamous cell skin cancer, in situ bladder cancer, or other cancer for which the patient has been disease-free for at least 2 years
16. Any other concurrent severe and/or uncontrolled concomitant medical condition that could compromise participation in the study (e.g., clinically significant pulmonary disease, clinically significant psychiatric or neurological disorder, active or uncontrolled infection)
17. Patient unwilling or unable to comply with this study protocol

PHASE 2

Phase 2 Inclusion Criteria

Patients must meet all of the following criteria to be enrolled in this study:

1. Age ≥ 18 years
2. ECOG Performance Status 0-1
3. Life expectancy of at least 12 weeks
4. Histologically or cytologically confirmed adenocarcinoma of the prostate (pure small cell carcinoma excluded)
5. Documented metastatic disease
6. Must have undergone bilateral orchiectomy (surgical castration) or willing to continue GnRH analog or antagonist (medical castration).
7. Serum testosterone <5 0 ng/dL
8. Progressive disease in the setting of medical or surgical castration (i.e., CRPC) as assessed by the investigator and that includes at least 1 of the following:

   1. Evidence of progression as measured by PSA defined as: PSA greater than or equal to 2 ng/mL (or PSA greater than or equal to 1 ng/mL if PSA progression is the only manifestation of progressive disease) and rising PSA by at least 2 consecutive measurements a minimum of 1-week apart and/or
   2. Soft tissue disease progression as per RECIST 1.1 and/or
   3. Bone disease progression defined by two or more new lesions on bone scan
9. Bisphosphonate or denosumab therapy allowed provided dose has been stable for ≥ 4 weeks prior to Day 1 of treatment.
10. Prior treatment:

    1. Only one prior line of a second-generation androgen inhibitor from a different class than the one chosen for the applicable phase 2 study (the 2 classes are CYP17 inhibitors [e.g., abiraterone, orteronel] and AR inhibitors [e.g., enzalutamide, apalutamide]). Patient must have progressed after ≥ 24 weeks of treatment with this second generation angrogen inhibitor
    2. No prior chemotherapy for mCRPC allowed; chemotherapy (including taxane-based) administered in the metastatic hormone-sensitive prostate cancer setting is allowed.
    3. Prior treatment with sipuleucel-T, radium-223, or other non-chemotherapy based treatments approved by the US FDA for the treatment of mCRPC is allowed; prior treatment with non-chemotherapy based treatments that are not approved for the treatment of mCRPC (e.g., pembrolizumab, ipilimumab, olaparib) are not allowed.
11. Recovery from recent surgery, radiotherapy, chemotherapy or other anti-cancer treatment to baseline or ≤ Grade 1 (other than alopecia)
12. Demonstrate adequate organ function
13. Patients who have not undergone a bilateral orchiectomy and have a female partner of childbearing potential must use an adequate barrier method of contraception during study treatment and for 90 days after receiving the last dose of CPI-1205 (or partner drug in the control arm of any randomized phase 2 trial if the patient does not participate in the crossover).
14. Willing to provide access to archival tumor tissue for research purposes, if available
15. Ability to swallow and retain oral medications.
16. Ability to understand and willingness to sign an IRB approved written ICF and authorization permitting release of personal health information including genetic testing relevant to cancer.
17. Able to comply with study visit schedule and assessments

Phase 2 Exclusion Criteria

Patients who meet any of the following criteria will not be enrolled in the study:

1. Known symptomatic brain metastases
2. Treatment with any of the following for prostate cancer within the indicated timeframe prior to Day 1 of treatment

   1. First-generation AR antagonists (e.g., bicalutamide, nilutamide, flutamide) within 4 weeks
   2. 5-alpha reductase inhibitors, ketoconazole, estrogens (including DES), or progesterones within 2 weeks
   3. Chemotherapy within 3 weeks
   4. Biologic therapy within 4 weeks
   5. Radionuclide therapy within 4 weeks
3. Radiation therapy for the treatment of metastasis within 1 week prior to Day 1 of treatment
4. Herbal products that may decrease PSA levels within 4 weeks prior to Day 1 of treatment
5. Systemic steroids > 10 mg of prednisone/prednisolone per day within 4 weeks prior to Day 1 of treatment
6. Major surgery within 4 weeks prior to Day 1 of treatment
7. Planned palliative procedures for alleviation of bone pain such as radiation therapy or surgery
8. Structurally unstable bone lesions concerning for impending fracture
9. Clinically significant cardiovascular disease including:

   1. MI/stroke within 6 months prior to day 1 of treatment
   2. Unstable angina within 3 months
   3. CHF with NYHA Class 3 or 4
   4. History of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsades de pointes)
   5. Uncontrolled hypertension (systolic BP > 170 mmHg or diastolic BP > 105 mmHg at screening) despite two concomitant antihypertensive therapies
   6. QTcF > 500 msec on the screening ECG
10. Active or symptomatic viral hepatitis or chronic liver disease
11. History of unresolved adrenal dysfunction
12. GI disorder that negatively affects absorption
13. Required treatment with one of the prohibited concomitant medications
14. Achlorhydria, either documented or suspected on the basis of an associated disease (e.g., pernicious anemia, atrophic gastritis, or certain gastric surgical procedures)
15. History of seizure, underlying brain injury with loss of consciousness, transient ischemic attack within 12 months prior to Day 1 of treatment, cerebral vascular accident or brain arteriovenous malformation
16. Known additional malignancy that is active and/or progressive requiring treatment; exceptions include basal cell or squamous cell skin cancer, in situ bladder cancer, or other cancer for which the patient has been disease-free for at least two years
17. Any other concurrent severe and/or uncontrolled concomitant medical condition that could compromise participation in the study (e.g., clinically significant pulmonary disease, clinically significant psychiatric or neurological disorder, active or uncontrolled infection)
18. Patient unwilling or unable to comply with this study protocol

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2021-02-03 (Actual); Study Completion 2021-02-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (41):
- United States (41):
  - Alaska Urological Institute, Anchorage, Alaska
  - Beverly Hills Cancer Center (BHCC), Beverly Hills, California
  - John Wayne Cancer Inst., Duarte, California
  - UCLA, Los Angeles, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - University of Colorado Hospital - Anschutz Cancer Pavilion, Aurora, Colorado
  - University of Florida, Jacksonville, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois Hospital and Health Systems, Chicago, Illinois
  - Indiana University- Simon Cancer Center, Indianapolis, Indiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - John Hopkins Kimmel Cancer Center, Baltimore, Maryland
  - Maryland Oncology Hematology, Rockville, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - GU Research Network, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - North Shore Hematology Oncology Associates, East Setauket, New York
  - NYU Langone Medical Center Laura and Isaac Permlutter Cancer Center, New York, New York
  - Icahn School of Medicine at Mt. Sinai, New York, New York
  - Eastchester Center for Cancer Care, The Bronx, New York
  - University of North Carolina-Chapel Hill, Chapel Hill, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University - James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - Toledo Clinic Cancer Center, Toledo, Ohio
  - Williamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Compass Oncology - East, Tualatin, Oregon
  - St. Luke's University, Bethlehem, Pennsylvania
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - Greenville Hospital System, Institute for Translational Oncology Research, Greenville, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Texas Oncology - Central Austin Cancer Center, Austin, Texas
  - Texas Oncology- Fort Worth, Fort Worth, Texas
  - Texas Oncology- Tyler, Tyler, Texas
  - Virginia Oncology Associates, Hampton, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1b Dose Escalation: CPI-1205 400 mg BID + Cobi + Enza: CPI-1205 400 mg BID in combination with Cobicistat 500 mg PO BID and Enzalutamide 160 mg PO QD
- Phase 1b Dose Escalation: CPI-1205 400 mg BID + Cobi + Abi/Pred: CPI-1205 400 mg BID in combination with Cobicistat 150 mg PO BID and Abiraterone 1000 mg PO QD and Prednisone 5 mg PO BID (28-day cycles)
- Phase 1b Dose Escalation: CPI-1205 800 mg TID + Enza: CPI-1205 800 mg TID in combination with Enzalutamide 160 mg PO QD (28-day cycles)
- Phase 1b Dose Escalation: CPI-1205 800 mg TID + Abi/Pred: CPI-1205 800 mg TID in combination with Abiraterone 1000 mg PO QD and Prednisone 5 mg PO BID (28-day cycles) Prednisone: Prednisone 5mg PO BID
- Phase 1b HPEC: CPI-1205 800 mg TID Heavily Pre-treated Expansion Cohort + Enza: CPI-1205 800 mg TID in heavily pretreated expansion cohort in combination with Enzalutamide 160 mg PO QD (28-day cycles)
- Phase 2 Randomized Controlled: Enza: Controlled group of Phase 2 randomized: Enzalutamide 160 mg PO QD
- Phase 2 Randomized Experimental: CPI-1205 at RP2D + Enza: CPI-1205 800 mg TID (RP2D) in combination with Enzalutamide 160 mg PO QD
- Phase 2 Single Arm: CPI-1205 (at RP2D) +Abi/Pred: CPI-1205 800 mg TID (RP2D) in combination with Abiraterone 1000 mg PO QD and Prednisone 5 mg PO BID (28-day cycles)
Period: Overall Study
Arm/Group | Phase 1b Dose Escalation: CPI-1205 400 mg BID + Cobi + Enza | Phase 1b Dose Escalation: CPI-1205 400 mg BID + Cobi + Abi/Pred | Phase 1b Dose Escalation: CPI-1205 800 mg TID + Enza | Phase 1b Dose Escalation: CPI-1205 800 mg TID + Abi/Pred | Phase 1b HPEC: CPI-1205 800 mg TID Heavily Pre-treated Expansion Cohort + Enza | Phase 2 Randomized Controlled: Enza | Phase 2 Randomized Experimental: CPI-1205 at RP2D + Enza | Phase 2 Single Arm: CPI-1205 (at RP2D) +Abi/Pred
Started (All enrolled patients) | 7 | 8 | 9 | 13 | 32 | 35 | 39 | 32
Phase 2: Crossover From Enza to CPI-1205 800mg TID + Enza (Crossed over patients from Enza alone arm to CPI-1205 800mg TID + Enza arm after progressing on Enza alone and having met the eligibility to participate in the cross-over arm and decision to initiate another systemic therapy for prostate cancer.) | 0 | 0 | 0 | 0 | 0 | 12 | 0 | 0
Safety Analysis Set (SAF) | 7 | 8 | 9 | 12 | 31 | 35 | 39 | 32
Full Analysis Set (FAS) | 7 | 8 | 9 | 12 | 31 | 35 | 39 | 32
Efficacy Analysis Set (EAS) | 5 | 7 | 9 | 11 | 25 | 35 | 38 | 28
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 8 | 9 | 13 | 32 | 35 | 39 | 32

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS)
Groups:
- Phase 1b Dose Escalation: CPI-1205 400 mg BID +Cobi + Enza: CPI-1205 400 mg BID in combination with Cobicistat 150mg PO BID and Enzalutamide 160 mg PO QD (28-day cycles)
- Phase 1b Dose Escalation: CPI-1205 400 mg BID + Cobi + Abi/Pred: CPI-1205 400 mg BID in combination iwth Cobicistat 150 mg PO BID and Abiraterone 1000 mg PO QD and Prednisone 5 mg PO BID (28-day cycles)
- Phase 1b Dose Escalation: CPI-1205 800 mg TID + Abi/Pred: CPI-1205 800 mg TID in combination with Abiraterone 1000 mg PO QD and Prednisone 5 mg PO BID (28-day cycles)
- Phase 1b HPEC: CPI-1205 800 mg TID Heavily Pretreated Expansion Cohort + Enza: CPI-1205 800 mg TID in heavily pretreated expansion cohort in combination with Enzalutamide 160 mg PO QD (28-day cycles)
- Phase 2 Randomized Controlled: Enza: Control group of Phase 2 randomized: Enzalutamide 160 mg PO QD
- Phase 2 Single Arm: CPI-1205 at RP2D + Abi/Pred: CPI-1205 800 mg TID (RP2D) in combination with Abiraterone 1000 mg PO QD and Prednisone 5 mg PO BID (28-day cycles)
- Total: Total of all reporting groups
Arm/Group | Phase 1b Dose Escalation: CPI-1205 400 mg BID +Cobi + Enza | Phase 1b Dose Escalation: CPI-1205 400 mg BID + Cobi + Abi/Pred | Phase 1b Dose Escalation: CPI-1205 800 mg TID + Enza | Phase 1b Dose Escalation: CPI-1205 800 mg TID + Abi/Pred | Phase 1b HPEC: CPI-1205 800 mg TID Heavily Pretreated Expansion Cohort + Enza | Phase 2 Randomized Controlled: Enza | Phase 2 Randomized Experimental: CPI-1205 at RP2D + Enza | Phase 2 Single Arm: CPI-1205 at RP2D + Abi/Pred | Total
Number analyzed (Participants) | 7 | 8 | 9 | 12 | 31 | 35 | 39 | 32 | 173
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 3 | 2 | 9 | 9 | 16 | 9 | 50
  >=65 years | 5 | 8 | 6 | 10 | 22 | 26 | 23 | 23 | 123
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 7 | 8 | 9 | 12 | 31 | 35 | 39 | 32 | 173
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 3 | 2 | 6 | 8 | 6 | 7 | 35
  White | 6 | 6 | 6 | 10 | 23 | 22 | 29 | 21 | 123
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 2 | 5 | 3 | 3 | 13
Prior cancer Immunotherapy [Count of Participants; unit: Participants] — Prior treatment received to enrollment
  Participants
    Yes | 2 | 4 | 4 | 4 | 14 | 8 | 10 | 12 | 58
    No | 5 | 4 | 5 | 8 | 17 | 27 | 29 | 20 | 115
Prior cancer hormonal Therapy [Count of Participants; unit: Participants] — Prior treatment received to enrollment
  Participants
    Yes | 7 | 8 | 9 | 12 | 31 | 35 | 39 | 31 | 172
    No | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Prior cancer chemotherapy [Count of Participants; unit: Participants] — Prior treatment received to enrollment
  Participants
    Yes | 3 | 3 | 3 | 4 | 31 | 7 | 9 | 8 | 68
    No | 4 | 5 | 6 | 8 | 0 | 28 | 30 | 24 | 105
Prior radiation therapy [Count of Participants; unit: Participants] — Prior treatment received to enrollment
  Participants
    Yes | 6 | 5 | 6 | 9 | 28 | 19 | 28 | 24 | 125
    No | 1 | 3 | 3 | 3 | 3 | 16 | 11 | 8 | 48

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Best Objective Response Rate Percent by Treatment Group
Description: Best overall response rate (%) defined as complete response (CR) + partial response (PR) divided by the total number of subjects as assessed by Investigator. The response assessment was performed per Prostate Cancer Working Group 3 (PCWG3) based on modifications of the RECIST 1.1 criteria. Per RECIST 1.1, a CR was assessed when all target lesions disappeared (any pathological lymph node must have reduction in short axis to <10 mm) in the post-baseline scan. A PR was assessed when there was at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 2 years [or until disease progression or unacceptable toxicity]
Population: Efficacy Analysis Set: subjects with a baseline measurement of response and at least 1 timepoint after baseline
Measure: Number (95% Confidence Interval); unit: Percent (%) of subjects
Groups:
- Phase 1b Dose Escalation: CPI-1205 400 mg BID + Cobi + Enza: CPI-1205 400 mg BID in combination with Cobicistat 150 mg PO BID and Enzalutamide 160mg PO QD (28-day cycles)
- Phase 1b Dose Escalation: CPI-1205 800 mg TID +Abi/Pred: CPI-1205 800 mg TID in combination with Abiraterone 1000 mg PO QD and Prednisone 5 mg PO BID (28-day cycles)
- Phase 1b HPEC: Heavily Pretreated Expansion Cohort CPI-1205 800 mg TID + Enza: Heavily pretreated expansion cohort (HPEC) CPI-1205 800 mg TID in combination with Enzalutamide 160mg PO QD (28-day cycles)
- Phase 2 Randomized Controlled: Enza: Phase 2 controlled group cohort randomized to Enzalutamide 160 mg PO QD (28-day cycles)
- Phase 2 Randomized Experimental: CPI-1205 at RP2D (800 mg TID) + Enza: CPI-1205 800 mg TID (RP2D) in combination with Enzalutamide 160 mg PO QD
- Phase 2 Randomized Crossover Period: CPI-1205 800 mg TID (RP2D) combination with Enzalutamide 160 mg PO QD
- Phase 2 Single Arm CPI-1205 at RP2D (800 mg TID) + Abi/Pred: CPI-1205 800 mg (RP2D) in combination with Abiraterone 1000 mg PO QD and Prednisone 5 mg PO BID (28-day cycles)
Arm/Group | Phase 1b Dose Escalation: CPI-1205 400 mg BID + Cobi + Enza | Phase 1b Dose Escalation: CPI-1205 400 mg BID + Cobi + Abi/Pred | Phase 1b Dose Escalation: CPI-1205 800 mg TID + Enza | Phase 1b Dose Escalation: CPI-1205 800 mg TID +Abi/Pred | Phase 1b HPEC: Heavily Pretreated Expansion Cohort CPI-1205 800 mg TID + Enza | Phase 2 Randomized Controlled: Enza | Phase 2 Randomized Experimental: CPI-1205 at RP2D (800 mg TID) + Enza | Phase 2 Randomized Crossover Period | Phase 2 Single Arm CPI-1205 at RP2D (800 mg TID) + Abi/Pred
Number analyzed (Participants) | 5 | 7 | 9 | 11 | 25 | 35 | 38 | 12 | 28
Percent (%) of subjects | 0 [0 to 52.18] | 0 [0 to 40.96] | 0 [0 to 33.63] | 0 [0 to 28.49] | 8.00 [0.98 to 26.03] | 5.71 [0.70 to 19.16] | 7.89 [1.66 to 21.38] | 0 [0 to 26.46] | 0 [0 to 12.34]

2. Primary Outcome: Efficacy: Percentage (%) of Subjects With PSA30
Description: The number of subjects who had a confirmed reduction of 30% of prostate-specific antigen (PSA30) from baseline
Time Frame: 2 years [or until progressive disease or unacceptable toxicity]
Population: Efficacy Analysis Set (EAS): Subset of Subjects with a baseline measurement PSA30 and at least 1 measurement post-baseline
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1b Dose Escalation: CPI-1205 400mg BID +Cobi+Enza: CPI-1205 Combination with Enzalutamide Drug: CPI-1205 PO 400mg BID OR Drug: CPI-1205 400mg BID/Cobicistat 150mg PO BID + Drug: Enzalutamide 160mg PO QD (28-day cycles) CPI-1205: CPI-1205 PO TID (either 400mg BID or 800mg TID during Phase 1 dose escalation study and at RP2D for Phase 2) Cobicistat: Cobicistat 150mg PO BID Enzalutamide: Enzalutamide 160mg PO QD
- Phase 1b Dose Escalation: CPI-1205 400mg BID +Cobi+Abi/Pred: CPI-1205 Combination with Abiraterone/Prednisone Drug: CPI-1205 PO 400mg BID OR Drug: CPI-1205 400mg BID/Cobicistat 150mg PO BID + Drug: Abiraterone 1000mg PO QD and 5mg Prednisone PO BID (28-day cycles) CPI-1205: CPI-1205 PO TID (either 400mg BID or 800mg TID during Phase 1 dose escalation study and at RP2D for Phase 2) Cobicistat: Cobicistat 150mg PO BID Abiraterone: Abiraterone 1000mg PO QD Prednisone: Prednisone 5mg PO BID
- Phase 1b Dose Escalation: CPI-1205 800mg TID +Enza; Phase 1b HPEC [Heavily Pre-treated Expansion Cohort] CPI-1205 800mg TID +Enza: CPI-1205 Combination with Enzalutamide Drug: CPI-1205 PO 800mg TID OR Drug: CPI-1205 800mg TID/Cobicistat 150mg PO BID + Drug: Enzalutamide 160mg PO QD (28-day cycles) CPI-1205: CPI-1205 PO TID (either 400mg BID or 800mg TID during Phase 1 dose escalation study and at RP2D for Phase 2) Cobicistat: Cobicistat 150mg PO BID Enzalutamide: Enzalutamide 160mg PO QD
- Phase 1b Dose Escalation: CPI-1205 800mg TID +Abi/Pred: CPI-1205 Combination with Abiraterone/Prednisone Drug: CPI-1205 PO 800mg TID OR Drug: CPI-1205 800mg TID/Cobicistat 150mg PO BID + Drug: Abiraterone 1000mg PO QD and 5mg Prednisone PO BID (28-day cycles) CPI-1205: CPI-1205 PO TID (either 400mg BID or 800mg TID during Phase 1 dose escalation study and at RP2D for Phase 2) Cobicistat: Cobicistat 150mg PO BID Abiraterone: Abiraterone 1000mg PO QD Prednisone: Prednisone 5mg PO BID
- Phase 2 Randomized Enza Contro: Enzalutamide Control Drug: Enzalutamide 160mg PO QD (28-day cycles) Enzalutamide: Enzalutamide 160mg PO QD
- Phase 2 Randomized Combination With Enza: CPI-1205 (at RP2D) Combination with Enzalutamide Drug: CPI-1205 (with or without cobicistat) at RP2D + Drug: Enzalutamide 160mg PO QD CPI-1205: CPI-1205 PO TID (either 400mg BID or 800mg TID during Phase 1 dose escalation study and at RP2D for Phase 2) Cobicistat: Cobicistat 150mg PO BID Enzalutamide: Enzalutamide 160mg PO QD
- Phase 2 Single Arm CPI-1205 +Abi/Pred: CPI-1205 (at RP2D) Combination with Abiraterone/Prednisone Drug: CPI-1205 (with or without cobicistat) at RP2D + Drug: Abiraterone 1000mg PO QD and Prednisone 5mg PO BID (28-day cycles) CPI-1205: CPI-1205 PO TID (either 400mg BID or 800mg TID during Phase 1 dose escalation study and at RP2D for Phase 2) Cobicistat: Cobicistat 150mg PO BID Abiraterone: Abiraterone 1000mg PO QD Prednisone: Prednisone 5mg PO BID
Arm/Group | Phase 1b Dose Escalation: CPI-1205 400mg BID +Cobi+Enza | Phase 1b Dose Escalation: CPI-1205 400mg BID +Cobi+Abi/Pred | Phase 1b Dose Escalation: CPI-1205 800mg TID +Enza | Phase 1b Dose Escalation: CPI-1205 800mg TID +Abi/Pred | Phase 1b HPEC [Heavily Pre-treated Expansion Cohort] CPI-1205 800mg TID +Enza | Phase 2 Randomized Enza Contro | Phase 2 Randomized Combination With Enza | Phase 2 Randomized Crossover Period | Phase 2 Single Arm CPI-1205 +Abi/Pred
Number analyzed (Participants) | 5 | 6 | 9 | 10 | 25 | 30 | 35 | 12 | 27
Participants | 1 | 1 | 2 | 1 | 7 | 7 | 12 | 1 | 4

3. Primary Outcome: Efficacy: Percentage (%) of Subjects With PSA50
Description: The number of subjects who had a confirmed reduction of 50% of prostate-specific antigen (PSA50) from baseline
Time Frame: 2 years [or until progressive disease or unacceptable toxicity]
Population: Efficacy Analysis Set (EAS): Subset of Subjects with a baseline measurement PSA50 and at least 1 measurement post-baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b Dose Escalation: CPI-1205 400mg BID +Cobi+Enza | Phase 1b Dose Escalation: CPI-1205 400mg BID +Cobi+Abi/Pred | Phase 1b Dose Escalation: CPI-1205 800mg TID +Enza | Phase 1b Dose Escalation: CPI-1205 800mg TID +Abi/Pred | Phase 1b HPEC [Heavily Pre-treated Expansion Cohort] CPI-1205 800mg TID +Enza | Phase 2 Randomized Enza Contro | Phase 2 Randomized Combination With Enza | Phase 2 Randomized Crossover Period | Phase 2 Single Arm CPI-1205 +Abi/Pred
Number analyzed (Participants) | 5 | 6 | 9 | 10 | 25 | 30 | 35 | 12 | 27
Participants | 1 | 1 | 1 | 1 | 4 | 5 | 10 | 0 | 2

4. Primary Outcome: Efficacy: Composite Response Rate (%) for Phase 2 Randomized and Phase 2 Single-arm Treatment Groups
Description: Subjects who had a circulating tumor cell of 30% (CTC 30%) or an objective response rate divided by the number of evaluable subjects
Time Frame: Up to 2 years [or until progressive disease or unacceptable toxicity]
Population: Efficacy Analysis Set (EAS): Subset of Subjects with an unfavorable assessment at baseline and at least one CTC assessment post baseline.
Measure: Number (95% Confidence Interval); unit: Percent (%) of subjects
Arm/Group | Phase 2 Randomized Enza Contro | Phase 2 Randomized Combination With Enza | Phase 2 Randomized Crossover Period | Phase 2 Single Arm CPI-1205 +Abi/Pred
Number analyzed (Participants) | 35 | 35 | 10 | 28
Percent (%) of subjects | 17.1 [6.6 to 33.6] | 31.4 [16.9 to 49.3] | 0 [0.0 to 30.8] | 21.4 [8.3 to 41.0]

5. Secondary Outcome: Efficacy: Best Responses by Treatment Group
Description: Best overall response defined as complete response (CR), partial response (PR); stable disease (SD); progressive disease (PD); and unknown/missing for the Phase 1b dose-escalation group, the Phase 1b HPEC group, the Phase 2 randomized groups, crossover group and the Phase 2 single-arm group. Assessed by Investigator
Time Frame: Up to 2 years [or until disease progression or unacceptable toxicity]
Population: Efficacy Analysis Set: subjects with a baseline measurement of response and at least 1 timepoint after baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b Dose Escalation: CPI-1205 400mg BID +Cobi+Enza | Phase 1b Dose Escalation: CPI-1205 400mg BID +Cobi+Abi/Pred | Phase 1b Dose Escalation: CPI-1205 800mg TID +Enza | Phase 1b Dose Escalation: CPI-1205 800mg TID +Abi/Pred | Phase 1b HPEC [Heavily Pre-treated Expansion Cohort] CPI-1205 800mg TID +Enza | Phase 2 Randomized Enza Contro | Phase 2 Randomized Combination With Enza | Phase 2 Randomized Crossover Period | Phase 2 Single Arm CPI-1205 +Abi/Pred
Number analyzed (Participants) | 5 | 7 | 9 | 11 | 25 | 35 | 38 | 12 | 28
Participants
  CR | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR | 0 | 0 | 0 | 0 | 2 | 2 | 3 | 0 | 0
  SD | 2 | 3 | 5 | 7 | 10 | 23 | 24 | 5 | 21
  PD | 3 | 3 | 4 | 1 | 10 | 9 | 7 | 0 | 5
  Not evaluable, unknown, or missing | 0 | 1 | 0 | 3 | 3 | 1 | 4 | 7 | 2

6. Secondary Outcome: Safety: Number of Participants With Treatment-emergent AEs Leading to Treatment Discontinuation
Description: Treatment-emergent Adverse events (AEs) leading to subjects withdrawing from treatment
Time Frame: Up to 2 years [or until clinical progression, radiographic disease progression, or until unacceptable toxicity]
Population: Safety Population: all subjects who receive any amount of treatment (includes phase Ib dose-escalation, phase 1b expansion, phase 2 randomized, phase 2 single-arm)
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b Dose Escalation: CPI-1205 400mg BID +Cobi+Enza | Phase 1b Dose Escalation: CPI-1205 400mg BID +Cobi+Abi/Pred | Phase 1b Dose Escalation: CPI-1205 800mg TID +Enza | Phase 1b Dose Escalation: CPI-1205 800mg TID +Abi/Pred | Phase 1b HPEC [Heavily Pre-treated Expansion Cohort] CPI-1205 800mg TID +Enza | Phase 2 Randomized Enza Contro | Phase 2 Randomized Combination With Enza | Phase 2 Randomized Crossover Period | Phase 2 Single Arm CPI-1205 +Abi/Pred
Number analyzed (Participants) | 7 | 8 | 9 | 12 | 31 | 35 | 39 | 12 | 32
Participants | 0 | 4 | 0 | 2 | 4 | 2 | 4 | 0 | 2

ADVERSE EVENTS:
Time Frame: Up to 2 years [or until progressive disease or unacceptable toxicity]
Groups:
- Phase 2 Randomized Control: Enza: Control group of Phase 2 randomized: Enzalutamide 160 mg PO QD (28-day cycles)
- Phase 2 Randomized Experimental: CPI-1205 at RP2D + Enza: CPI-1205 800 mg TID (RP2D) in combination with Enzalutamide 160 mg PO QD (28-day cycles)
- Phase 2 Single Arm: CPI-1205 (at RP2D) + Abi/Pred: CPI-1205 800 mg TID (RP2D) in combination with Abiraterone 1000 mg PO QD and Prednisone 5 mg PO BID (28-day cycles)
Arm/Group | Phase 1b Dose Escalation: CPI-1205 400 mg BID + Cobi + Enza | Phase 1b Dose Escalation: CPI-1205 400 mg BID + Cobi + Abi/Pred | Phase 1b Dose Escalation: CPI-1205 800 mg TID + Enza | Phase 1b Dose Escalation: CPI-1205 800 mg TID + Abi/Pred | Phase 1b HPEC: CPI-1205 800 mg TID Heavily Pretreated Expansion Cohort + Enza | Phase 2 Randomized Control: Enza | Phase 2 Randomized Experimental: CPI-1205 at RP2D + Enza | Phase 2 Randomized Crossover Period | Phase 2 Single Arm: CPI-1205 (at RP2D) + Abi/Pred
All-Cause Mortality (participants affected / at risk) | 1/7 | 2/8 | 1/9 | 1/12 | 17/31 | 10/35 | 7/39 | 4/12 | 9/32
Serious Adverse Events (participants affected / at risk) | 2/7 | 3/8 | 2/9 | 1/12 | 11/31 | 8/35 | 5/39 | 0/12 | 1/32
Other Adverse Events (participants affected / at risk) | 7/7 | 8/8 | 9/9 | 12/12 | 31/31 | 33/35 | 38/39 | 11/12 | 30/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b Dose Escalation: CPI-1205 400 mg BID + Cobi + Enza (N=7) | Phase 1b Dose Escalation: CPI-1205 400 mg BID + Cobi + Abi/Pred (N=8) | Phase 1b Dose Escalation: CPI-1205 800 mg TID + Enza (N=9) | Phase 1b Dose Escalation: CPI-1205 800 mg TID + Abi/Pred (N=12) | Phase 1b HPEC: CPI-1205 800 mg TID Heavily Pretreated Expansion Cohort + Enza (N=31) | Phase 2 Randomized Control: Enza (N=35) | Phase 2 Randomized Experimental: CPI-1205 at RP2D + Enza (N=39) | Phase 2 Randomized Crossover Period (N=12) | Phase 2 Single Arm: CPI-1205 (at RP2D) + Abi/Pred (N=32)
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0
Pelvic mass (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | NA | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | NA | 0
Anal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | NA | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | NA | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | NA | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | NA | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | 0
Cellullitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | 0
Streptococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | 0
Musculoskeletal procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b Dose Escalation: CPI-1205 400 mg BID + Cobi + Enza (N=7) | Phase 1b Dose Escalation: CPI-1205 400 mg BID + Cobi + Abi/Pred (N=8) | Phase 1b Dose Escalation: CPI-1205 800 mg TID + Enza (N=9) | Phase 1b Dose Escalation: CPI-1205 800 mg TID + Abi/Pred (N=12) | Phase 1b HPEC: CPI-1205 800 mg TID Heavily Pretreated Expansion Cohort + Enza (N=31) | Phase 2 Randomized Control: Enza (N=35) | Phase 2 Randomized Experimental: CPI-1205 at RP2D + Enza (N=39) | Phase 2 Randomized Crossover Period (N=12) | Phase 2 Single Arm: CPI-1205 (at RP2D) + Abi/Pred (N=32)
Fatigue (General disorders) | 3 | 3 | 7 | 4 | 12 | 18 | 23 | 6 | 6
Axillary Pain (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Peripheral edema (General disorders) | 2 | 0 | 2 | 2 | 2 | 2 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 6 | 5 | 14 | 6 | 21 | 8 | 18
Nausea (Gastrointestinal disorders) | 0 | 3 | 5 | 4 | 15 | 6 | 12 | 4 | 9
Constipation (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 7 | 3 | 4 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 3 | 3 | 2 | 1 | 3
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 5 | 2 | 9 | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1 | 3 | 6 | 9 | 3 | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 4 | 2 | 5 | 5 | 5 | 2 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1 | 5 | 3 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 4 | 0 | 1 | 7 | 1 | 6
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3 | 2 | 3 | 9 | 5 | 9 | 1 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 2 | 2 | 3 | 2 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 3 | 2 | 0 | 1 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 2 | 1 | 1 | 0 | 2
Headache (Nervous system disorders) | 0 | 1 | 2 | 3 | 2 | 1 | 6 | 0 | 2
Dizziness (Nervous system disorders) | 1 | 2 | 2 | 1 | 5 | 0 | 2 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 1 | 0 | 5 | 3 | 4 | 2 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 1 | 0 | 1 | 0 | 4 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 2 | 1 | 0 | 1 | 0 | 3 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 2 | 4 | 4 | 1 | 2
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 3 | 5 | 5 | 4 | 4 | 6
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 2 | 4 | 3 | 0 | 1 | 2
Hematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 3 | 4 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-07-26): https://cdn.clinicaltrials.gov/large-docs/46/NCT03480646/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-13): https://cdn.clinicaltrials.gov/large-docs/46/NCT03480646/SAP_001.pdf